CLINICAL TRIAL: NCT07247266
Title: A Phase 1b, Open-label, Single-arm Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of JTE-162 in Subjects With Cryopyrin-Associated Periodic Syndrome (CAPS)
Brief Title: Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of JTE-162 in Subjects With Cryopyrin-Associated Periodic Syndrome (CAPS)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AE162-X-24-003
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Cryopyrin-associated Periodic Syndromes (CAPS)
Keywords: JTE-162; Efficacy; Safety; Tolerability; Cryopyrin-associated periodic syndromes; CAPS; Pharmacokinetics
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JTE-162 Tablets (Experimental): Dose 1 once daily for 2 Weeks
  Interventions: Drug: JTE-162

INTERVENTIONS:
Drug: JTE-162 — Tablets containing JTE-162

SUMMARY:
This study will evaluate the efficacy, safety, tolerability and pharmacokinetics of JTE-162 administered once daily for 2 weeks in subjects with cryopyrin-associated periodic syndrome (CAPS)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with familial cold autoinflammatory syndrome (FCAS) or Muckle-Wells syndrome (MWS) confirmed by:
* Clinical History: At least 2 typical clinical symptoms (e.g., urticarial skin rash, myalgia, arthralgia, recurrent fever, fatigue/malaise, conjunctivitis or other autoinflammatory symptoms) prior to the Screening Visit; AND
* Genetic Confirmation: Confirmed nucleotide-binding and oligomerization domain (NOD)-like receptor family pyrin domain containing 3 (NLRP3) mutation;
* Willing to discontinue current anti-interleukin (IL)-1 treatment, if applicable;
* Demonstrates de novo flaring of CAPS during the Screening Period.

Exclusion Criteria:

* Has chronic infantile neurologic cutaneous articular syndrome (CINCA)/neonatal-onset multisystem inflammatory disease (NOMID);
* Has a history or presence of amyloidosis, progressive hearing loss, organ damage or any symptom contraindicating anti-IL-1 treatment washout;
* Has active systemic bacterial, fungal or viral infection(s) within 14 days prior to Day 1 or a history of clinically significant recurrent infectious diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change and percent change from baseline to end of treatment (EOT) in high-sensitivity C-reactive protein (hs-CRP) | 2 Weeks
Change and percent change from baseline to EOT in Serum amyloid A (SAA) | 2 Weeks
Change and percent change from baseline to EOT in Interleukin (IL)-6 | 2 Weeks
Change and percent change from baseline to EOT in Key symptom score (KSS) | 2 Weeks
Change and percent change from baseline to EOT in Individual symptom score on Daily Health Assessment Form, Second Generation (DHAF2) | 2 Weeks
Change and percent change from baseline to EOT in Global assessments of disease activity on DHAF2 | 2 Weeks
Change and percent change from baseline to EOT in Global CAPS symptom assessment by the Investigator | 2 Weeks
Change and percent change from baseline to EOT in Individual CAPS symptom assessment by the Investigator | 2 Weeks
Number of adverse events | 4 Weeks
JTE-162 post-dose plasma concentrations on Day 1 | 1 Day
JTE-162 trough plasma concentrations on Days 2, 3 and 4, and at the Week 2 Visit (Day 15±2) | Day 2, Day 3, Day 4 and Day 15±2

CONTACTS AND LOCATIONS:
Locations (1):
- Gordon Sussman Clinical Research Inc., North York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No